CLINICAL TRIAL: NCT00298636
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Escalating Dose-Response Trial of Intravenous Adenosine for Perioperative Analgesia in Females Undergoing Abdominal Hysterectomy or Myomectomy
Brief Title: Dose-Response of Adenosine for Perioperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xsira Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ADO-122
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-08

CONDITIONS: Perioperative Pain
MeSH Terms: interventions — Adenosine

INTERVENTIONS:
Drug: adenosine

SUMMARY:
Adenosine A1 and A2 receptors are widely distributed in the brain and spinal cord and represent a non-opiate target for pain management. Activated spinal A1 receptors inhibit sensory transmission by inhibiting the slow ventral root potential, which is the C-fiber-evoked excitatory response associated with nociception. Adenosine may inhibit intrinsic neurons through an increase in K+ conductance and presynaptic inhibition of sensory nerve terminals to inhibit the release of substance P and perhaps glutamate. Although adenosine A3 receptors are not found in the nervous system, adenosine is also known to have anti-inflammatory properties that may contribute to pain relief in the peripheral setting of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Female gender; age 18 to 65 years;
* American Society of Anesthesiology (ASA) physical classification I to III;
* scheduled for non-emergent abdominal hysterectomy (with or without salpingo-oophorectomy) or myomectomy under general anesthesia;

Exclusion Criteria:

* ASA physical classification of IV or V;
* documented history of cardiovascular disease including coronary artery disease, uncontrolled hypertension, aortic stenosis, congestive heart failure, cardiac arrhythmias or conduction defects greater that first degree atrioventricular (AV) block, sinoatrial (SA) or AV node disease including sick sinus syndrome or symptomatic bradycardia, presence of devices including pacemakers or internal defibrillators, or history of symptoms consistent with any of the aforementioned conditions (e.g., angina, dyspnea on exertion, paroxysmal nocturnal dyspnea);
* history of asthma, bronchospastic lung disease, or hyper-reactive airway disease;
* history of gout;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-10

PRIMARY OUTCOMES:
Dose-response

SECONDARY OUTCOMES:
efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Tong J Gan, M.D., Principal Investigator — Duke University
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - University of Miami/Miller School of Medicine, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University/Forsyth Medical Center, Winston-Salem, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Memorial Hermann-Memorial City Hospital, Houston, Texas